CLINICAL TRIAL: NCT03640104
Title: Effect of an Individualized Dietary Intervention on the Body Composition and Vitamin A Status of Breastfeeding Women
Brief Title: Individualized Dietary Intervention in Breastfeeding Women: Body Weight and Vitamin A Stores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Sonora (Other)
Collaborators: Centro de Investigación en Alimentación y Desarrollo A.C. (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Verónica López Teros, PhD, Research professor, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLT-001
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Overweight and Obesity; Vitamin A Deficiency; Dietary Modification; Breastfeeding
Keywords: Food-based intervention; postpartum weight management; hepatic retinol
MeSH Terms: conditions — Overweight; Obesity; Vitamin A Deficiency; Breast Feeding | interventions — Nutrition Policy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Nutrition guidelines (Experimental): Subjects will receive an individualized dietary plan according to their nutritional status, socioeconomic and cultural preferences. Protein intake 1-1.5g/kg body weight; 30% fat (mono and polyunsaturated fatty acids), vitamin A sources (1300 RAE). Each subject will have 7 interchangeable options for every meal time, all equivalent in macronutrient content, and every two weeks a new menu will be provided by a nutritionist.
  Interventions: Behavioral: Intervention-Nutrition guidelines
- Nutrition Guidelines (Other): Participants will receive general nutritional recommendations according to international standards
  Interventions: Behavioral: Nutrition guidelines

INTERVENTIONS:
Behavioral: Intervention-Nutrition guidelines — Subjects will receive an individualized dietary plan according to their nutritional status, socioeconomic and cultural preferences. Protein intake 1-1.5g/kg body weight; 30% fat (mono and polyunsaturated fatty acids), vitamin A sources (1300 RAE). Each subject will have 7 interchangeable options for every meal time, all equivalent in macronutrient content, and every two weeks a new menu will be provided by a nutritionist.
  Arms: Intervention-Nutrition guidelines
Behavioral: Nutrition guidelines — Nutritional recommendations based on international guidelines
  Arms: Nutrition Guidelines

SUMMARY:
Breast milk is the best food during the first 6mo of life because it offers multiple benefits for the mother-infant pair. An inadequate maternal diet during pregnancy can lead to excess weight gain, leading to negative health consequences for the dyad. In Mexico, an excess of body weight coexists with micronutrient deficiencies (double burden of malnutrition). Low vitamin A concentration has been observed in northwest Mexico, which can affect the human milk composition and increase the risk of VAD in breastfed babies. An individualized dietary intervention in the lactating woman will reduce body weight and improve vitamin A status. The objective is to assess the effect of an individualized dietary intervention during 3 months postpartum on body composition and vitamin A status of lactating women.

DETAILED DESCRIPTION:
This protocol was approved by the Bioethics Committee of the Department of Medicine and Health Sciences of Universidad de Sonora. A randomized controlled trial will be carried out and participant women will be assigned by simple randomization 1:1 to either the intervention or control group, upon signing an informed consent. At baseline (2wk postpartum), anthropometric (weight, height, mid upper-arm circumference and triceps skinfold thickness) and body composition (DXA) measurements as well as the assessment of vitamin A status (serum and breastmilk retinol and the modified relative dose response) will be performed. The control group will receive only recommendations for a healthy diet in accordance with international standards and will be followed up every month to promote adherence and to assess their nutritional status. On the other hand, the intervention group will receive an individualized macronutrient meal equivalent menu, with nutritional consultations every two weeks. The dietary plan will include 1-1.5 g/kg body weight protein, 30% total fat (preferably mono and polyunsaturated fatty acids), and vitamin A sources (1300 RAE). After 3 months of intervention are completed, baseline measurements will be repeated. Statistical analysis will include descriptive stats and comparisons between groups (t-tests), significance will be defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25
* Predominant breastfeeding
* Signed Informed Consent

Exclusion Criteria:

* Multiparity
* Alcohol, drugs, tobacco intake
* Use of dietary supplements
* Active infection (C reactive protein > 6mg/L)
* External nutritional counseling
* Pregnancy during the study period
* Liver disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Total Body weight | Baseline and 3 months after enrollment
  Difference in change (between baseline and final body weight within groups) between the intervention and control group, respectively
Vitamin A liver stores | Baseline and 3 months after enrollment
  Stores are calculated as the DR/R ratio. The outcome will be calculated as the difference in change (between baseline and final VA stores within groups) between the intervention and control group, respectively

SECONDARY OUTCOMES:
Body fat mass | Baseline and 3 months after enrollment
  Difference in change (between baseline and final body fat mass within groups) between the intervention and control group, respectively
Retinol | Baseline and 3 months after enrollment
  Difference in change (between baseline and final retinol concentration within groups) between the intervention and control group, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Lopez-Teros, Dr, Principal Investigator — Universidad de Sonora
Locations (1):
- Universidad de Sonora, Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No